CLINICAL TRIAL: NCT05597553
Title: Clinical and Radiographic Evaluation of Premixed Verses Powder / Liquid Bioceramic Mineral Trioxide Aggregate in Indirect Pulp Capping of Immature Permanent Mandibular Molars: A Randomized Clinical Trial
Brief Title: Evaluation of Premixed Verses Powder/Liquid Bioceramic MTA in Indirect Pulp Capping.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aisha Magdy Khairy Abozaid, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PM Mta verses P/L
Record Dates: First submitted 2022-10-19; First posted 2022-10-28 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Indirect Pulp Capping
MeSH Terms: interventions — Powders

STUDY DESIGN:
Intervention Model Description: Mineral trioxide aggregate (MTA) is a bioactive, biocompatible, antibacterial material with good stability and excellent sealing ability that has been used as a dressing material in pulp capping procedures in permanent teeth
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premixed MTA (Experimental): The premixed bioceramics putty are ready to use materials, fast setting, with superior handling properties and hydrophilic in nature that necessitate moisture from the adjacent tissues to set. They have advantage of insensitive to moisture and blood contamination with less technique sensitive.
  Interventions: Other: Premixed MTA; Other: Powder/liquid MTA
- Powder/liquid MTA (Active Comparator): Mineral trioxide aggregate (MTA) is a bioactive, biocompatible, antibacterial material with good stability, and excellent sealing ability that has been used as a dressing material in pulp capping procedures in permanent teeth, although it has good properties, it has many limitations, including long setting time, handling property and tooth discoloration making the use of this material challenging for many clinicians.
  Interventions: Other: Premixed MTA; Other: Powder/liquid MTA

INTERVENTIONS:
Other: Premixed MTA — The premixed Bio-ceramic putty during setting become hard and expand slightly providing a superior long-term seal
  Other Names: MTA Putty
Other: Powder/liquid MTA — Mineral trioxide aggregate (MTA) is a silicate material that is said to aid in faster bridge formation with fewer tunnel defects, less pulpal inflammation, and the maintenance of pulpal integrity. It is widely used in pediatric dentistry due to its excellent sealing properties.

SUMMARY:
Evaluate Clinical and Radiographic Evaluation of Premixed verses Powder / Liquid Bioceramic Mineral Trioxide Aggregate in Indirect Pulp Capping of Immature Permanent Mandibular Molars

DETAILED DESCRIPTION:
Mineral trioxide aggregate (MTA) is a bioactive, biocompatible, antibacterial material with good stability, and excellent sealing ability that has been used as a dressing material in pulp capping procedures in permanent teeth.

Although it has good properties, MTA has many limitations, including long setting time, handling property and tooth discoloration making the use of this material challenging for many clinicians.

Researchers and manufacturers have made progress in overcoming these problems in recent years, new and improved products are becoming available such as the premixed bioceramic putty.

The premixed bioceramics putty are ready to use materials, fast setting, with superior handling properties and hydrophilic in nature that necessitate moisture from the adjacent tissues to set. They have advantage of insensitive to moisture and blood contamination with less technique sensitive. Upon setting, they become hard and expand slightly providing with superior long-term seal.

Premixed Bio-ceramics (BC) are highly alkaline materials (pH = 12.7), they release calcium and have antibacterial activity. Their biocompatibility is higher than that of MTA, this is attributed to the absence of heavy metals from the premixed BC components.

The premixed bio-ceramic putty (Well-Root™ PT) has been developed for the management of pulp capping procedures with the advantage of uniform homogenous consistency and lack of waste. It is radiopaque material based on a calcium aluminosilicate composition.

It has excellent biological & physical properties and does not shrink during setting. Well-Root™ PT does not create an inflammatory response and promotes mineralization.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit and cooperative children.
* Pediatric patients aged 6-8 years.
* Deep caries with reversible pulpits in immature first permanent mandibular molars indicated for indirect pulp capping.
* Absence of clinical signs and symptoms of pulpal exposure.
* Absence of radiographic signs and symptoms of pulp degeneration.
* Positive parental informed consent.

Exclusion Criteria:

* Clinical symptoms of irreversible pulpitis requiring endodontic treatment.
* Clinical symptoms of pulp exposure.
* The presence of fistulas or swelling.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 12months
  Clinical examination by(Visual Analogue Scale) System (0 - Mild - Moderate - Severe)

SECONDARY OUTCOMES:
Pulp vitality | 12months
  Evaluate of pulp vitality by Electrical pulp test 9Normal response, Exaggerated brief Exaggerated prolong, Negative)
Absence of furcal radiolucency or root resorption | 12months
  Evaluate Periapical Intraoral Digital Radiography if present or absent

CONTACTS AND LOCATIONS:
Overall Officials: Mai Mohamed, Lecturer, Study Director — Cairo University

REFERENCES:
- [Result] Torabinejad M, Parirokh M, Dummer PMH. Mineral trioxide aggregate and other bioactive endodontic cements: an updated overview - part II: other clinical applications and complications. Int Endod J. 2018 Mar;51(3):284-317. doi: 10.1111/iej.12843. Epub 2017 Oct 11. PMID 28846134
- [Result] Abdelmotelb MA, Gomaa YF, Khattab NMA, Elheeny AAH. Premixed bioceramics versus mineral trioxide aggregate in furcal perforation repair of primary molars: in vitro and in vivo study. Clin Oral Investig. 2021 Aug;25(8):4915-4925. doi: 10.1007/s00784-021-03800-3. Epub 2021 Jan 22. PMID 33483869
- [Result] Motwani N, Ikhar A, Nikhade P, Chandak M, Rathi S, Dugar M, Rajnekar R. Premixed bioceramics: A novel pulp capping agent. J Conserv Dent. 2021 Mar-Apr;24(2):124-129. doi: 10.4103/JCD.JCD_202_20. Epub 2021 Oct 9. PMID 34759576